CLINICAL TRIAL: NCT00952601
Title: Pilot Study of the Modified Atkins Diet for Tourette Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient interest and recruitment - study ended prematurely by investigators
Sponsor: Johns Hopkins University (Other)
Responsible Party: Eric Kossoff MD, Johns Hopkins University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AtkinsTourette
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Tourette Syndrome
Keywords: Tourette; Atkins; Ketosis; Tic
MeSH Terms: conditions — Tourette Syndrome; Ketosis; Tics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modified Atkins Diet (Experimental): Patients are started on the modified Atkins diet at 15 grams per day.
  Interventions: Dietary Supplement: Modified Atkins diet

INTERVENTIONS:
Dietary Supplement: Modified Atkins diet — Low carbohydrate diet

SUMMARY:
Pharmacotherapy has long been considered the primary approach for tic suppression in Tourette syndrome (TS). Unfortunately, medications are often ineffective and frequently have significant side-effects. This is a pilot therapeutic study using a dietary approach, the modified Atkins diet (MAD). The goal of this study is to establish the safety, tolerability, and efficacy of dietary therapy in patients with TS ("proof of concept") and to determine whether this intervention is worthy of evaluation in large-scale clinical trials. The modified Atkins diet mimics the well established ketogenic diet, but in a less-restrictive dietary manner. Dietary approaches using the MAD/ketogenic diet are currently under investigation for neurological conditions other than epilepsy, including Alzheimer disease, headaches, autism, narcolepsy, brain tumors, traumatic brain injury, Parkinson's disease, and depression.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-65 years
* Tourette syndrome (vocal and motor tics for over a year)
* > 20 score on the Yale Global Tic Severity Scale
* Ability to follow instructions and comply with the dietary changes

Exclusion Criteria:

* Secondary tics
* Underweight (BMI < 5%)
* Prior use of the Atkins diet for over 2 days
* High cholesterol or triglycerides
* Major depression or anxiety disorder
* Pregnancy
* Substance abuse

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Tic frequency | 2 months
  Number of tics per day, intensity, severity, will be compared to baseline (pre-diet)

SECONDARY OUTCOMES:
Ketosis | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kossoff EH, Dorward JL. The modified Atkins diet. Epilepsia. 2008 Nov;49 Suppl 8:37-41. doi: 10.1111/j.1528-1167.2008.01831.x. PMID 19049584